CLINICAL TRIAL: NCT04975659
Title: Placebo Versus Nocebo: Effects on Pain and Anxiety During Local Anaesthetic Infiltration in Parturient Undergoing Elective Caesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Kebangsaan Malaysia Medical Centre (Other)
Responsible Party: Principal Investigator, Rufinah Teo, Lecturer and Consultant Anesthesiologist , Department of Anesthesia and Intensive Care, Universiti Kebangsaan Malaysia Medical Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UKM PPl/111/8/JEP-2020-011
Record Dates: First submitted 2021-07-02; First posted 2021-07-23 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Communication
Keywords: Placebo; Nocebo; Pain; Anxiety; Local Skin Infiltration
MeSH Terms: conditions — Communication; Pain; Anxiety Disorders | interventions — Nocebo Effect

STUDY DESIGN:
Intervention Model Description: We randomised participants into either the nocebo (N) or placebo (P) group using computer generated numbers
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants are blinded from their randomization. Personnel assessing the pain score is blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nocebo (Active Comparator): We informed subjects in the N group a negative suggestion, using the following script: "During the local anaesthetic injection, you are going to feel a sharp prick at your back; this is usually the painful part of the procedure"
  Interventions: Behavioral: Placebo and Nocebo effect
- Placebo (Placebo Comparator): We informed subjects in the P group a positive suggestion, using the following script: "We will administer some local anaesthetic to numb your back; this will allow the procedure to be more comfortable and tolerable for you."
  Interventions: Behavioral: Placebo and Nocebo effect

INTERVENTIONS:
Behavioral: Placebo and Nocebo effect — Positive suggestion and words is used on Placebo group Negative suggestion and words is used on Nocebo group

SUMMARY:
This randomized trial compared placebo and nocebo effect over anaesthetist-patient communication on pain and anxiety score during local anaesthetic (LA) skin infiltration in parturient undergoing caesarean delivery under regional anaesthesia (RA). A secondary objective was to determine if education level and previous RA experience affect pain and anxiety scores. Parturients scheduled for elective caesarean delivery were randomised into Placebo (P) or Nocebo (N) group. Baseline Amsterdam Preoperative Anxiety & Information Scale (APAIS0) were obtained. Standardised scripts describing the LA skin infiltration for RA were used during the pre-anaesthetic review. (N) group were explained with words like "pain, prick, sharp" while words like "numb, comfort, tolerable" were used in the (P) group, avoiding "painful" expressions. The same scripts will be repeated before skin infiltration during the RA procedure. On the day of surgery, a second (APAIS1) was obtained upon arrival to the theatre. Pain score using the numerical rating scale (NRS) was assessed after LA infiltration.

DETAILED DESCRIPTION:
We randomised participants into either the nocebo (N) or placebo (P) group. We obtained a baseline anxiety score (APAIS0) using the Amsterdam Preoperative Anxiety and Information Scale (APAIS) during the pre-anaesthesia visit. Following that, we informed subjects in the N group a negative suggestion, using the following script: "During the local anaesthetic injection, you are going to feel a sharp prick at your back; this is usually the most painful part of the procedure". On the other hand, we used a positive suggestion on the P group: "We will administer some local anaesthetic to numb your back; this will allow the procedure to be more comfortable and tolerable for you." We obtain a second anxiety score (APAIS1) in the operating theatre before the caesarean section. We carried out either spinal anaesthesia or continuous spinal epidural according to standard hospital protocol and indication. Before the LA skin infiltration, the anaesthetist repeats the same script to the subjects according to the prior randomisation. Five millilitres of lignocaine 2% is injected intradermally and subcutaneously by the anaesthetist into interspinous space in a single pass through a 22-gauge needle to create a skin wheal.

During the LA infiltration, only the attending anaesthetist performing the procedure gave participants verbal instructions; other personnel remained silent throughout. We recorded the presence of vocalisation of pain, withdrawal movement or facial grimacing. Immediately after the LA infiltration, a blinded and trained general anaesthetic nurse or personnel enters the operating theatre to assess the subjects' pain score using the numerical rating scale (NRS). After collection of the pain score, the anaesthetist performed the remaining anaesthetic procedure as per clinical routine.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiology (ASA) II category parturient listed for elective caesarean delivery.
* Can understand intended verbal communication

Exclusion Criteria:

* receiving any form of analgesia within 6 hours before the study
* chronic pain,
* anxiety disorders
* allergy to Local Anaesthetic drugs

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Actual)
Dates: Start 2020-07-13 (Actual); Primary Completion 2021-05-21 (Actual); Study Completion 2021-05-28 (Actual)

PRIMARY OUTCOMES:
Pain score | Throughout study completion, average of 10 months
  Pain score during local anaesthetic infiltration using Numerical Rating Scale (NRS) (range 0-10) where 0 is "no pain at all" and 10 is " worst pain ever felt"
Baseline anxiety score | Through study completion, average of 10 months
  Validated questionnare using the Amsterdam Preoperative Anxiety & Information Scale. (APAIS) (Range 6-30). Higher scores mean higher anxiety level
Preoperative anxiety score | Through study completion, average of 10 months
  Validated questionnare using the Amsterdam Preoperative Anxiety & Information Scale. (Range 6-30). Higher scores mean higher anxiety level

SECONDARY OUTCOMES:
Association of Education level on Pain and anxiety score | Through study completion, average of 10 months
  Correlation between subjects education level on pain score (NRS) and anxiety score (APAIS)
Association of past history of regional anesthesia on Pain and anxiety score | Through study completion, average of 10 months
  Correlation between subjects previous experience of regional anesthesia on pain score (NRS) and anxiety score (APAIS)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz,, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mohd Fahmi Z, Lai LL, Loh PS. Validation of the Malay version of the Amsterdam Preoperative Anxiety and Information Scale (APAIS). Med J Malaysia. 2015 Aug;70(4):243-8. PMID 26358022
- [Background] Dutt-Gupta J, Bown T, Cyna AM. Effect of communication on pain during intravenous cannulation: a randomized controlled trial. Br J Anaesth. 2007 Dec;99(6):871-5. doi: 10.1093/bja/aem308. Epub 2007 Oct 30. PMID 17977860
- [Result] Varelmann D, Pancaro C, Cappiello EC, Camann WR. Nocebo-induced hyperalgesia during local anesthetic injection. Anesth Analg. 2010 Mar 1;110(3):868-70. doi: 10.1213/ANE.0b013e3181cc5727. Epub 2009 Dec 30. PMID 20042440
- [Result] Moerman N, van Dam FS, Muller MJ, Oosting H. The Amsterdam Preoperative Anxiety and Information Scale (APAIS). Anesth Analg. 1996 Mar;82(3):445-51. doi: 10.1097/00000539-199603000-00002. PMID 8623940